CLINICAL TRIAL: NCT04252807
Title: Evaluating the Impact of a Common Elements-based Intervention to Improve Maternal Psychological Well-being and Mother-infant Interaction in a Low Resource Community Setting of Rural Pakistan
Brief Title: A Common Elements-based Intervention to Improve Maternal Psychological Well-being and Mother-infant Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: World Health Organization (Other); University of Liverpool (Other); Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCC definitive cRCT
Record Dates: First submitted 2019-09-14; First posted 2020-02-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Maternal Distress; Perinatal Depression; Development Delay; Language Delay; Cognitive Developmental Delay; Nutrition Poor; Growth Delay; Motor Delay; Maternal Behavior; Infant Development; Infant Malnutrition; Infant Behavior
MeSH Terms: conditions — Learning Disabilities; Language Development Disorders; Malnutrition; Psychomotor Disorders; Infant Nutrition Disorders; Infant Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Single blind, two arm, individual randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators and outcome assessors will be blind to the allocations status of participants. To ensure blinding, participants will be instructed to not disclose their allocation during assessment.
  Fidelity of masking will be ensured by having assessors guess the allocation status of participants at the end of assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Distressed mothers randomized to intervention arm will receive a common elements based integrated intervention that combines evidence based elements from packages of care addressing early stimulation, responsive feeding and perinatal depression. The integrated intervention is expected to a) improve mother psychological distress, b) improve family support, c) improve child development and d) promote mother-infant interaction.
  The participants will receive 15 monthly sessions at home by lay health workers. First three sessions will be delivered to the participants in the third trimester of pregnancy, followed by 12 monthly sessions afterwards.
  Interventions: Behavioral: Intervention arm
- Treatment as Usual (TAU) (Active Comparator): The participants in the control arm will receive the routine monthly visits by the trained Lady Health Workers (LHWs) of their respective areas.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Intervention arm — In addition to the routine care delivered by Lady Health Workers (LHWs), the participants in the intervention arm will receive common elements based integrated intervention. The providers of the intervention are lay health workers who will be trained in the intervention using an online course. The lay health worker will complete the online training course in a group, with interactive group activities and role plays. Lay health workers will be supported online and in-person by the trainers in monthly supervision meetings. The lay health workers will deliver intervention to distressed mothers in 15 monthly sessions. The intervention consists of three modules including 1) mothers' well-being, 2) infant nutrition,early stimulation and breastfeeding and 3) mother-infant interaction.
  Arms: Intervention arm
Other: Treatment as Usual — The participants in the control arm will receive the routine visits by LHWs of their respective areas. The LHWs are trained to provide antenatal care and referral, immunization services and support to community mobilization, provision of family planning and basic curative care via door to door visits to the households of their allocated areas.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Background: Millions of children in low resource settings are at high risk of poor development due to factors such as undernutrition, inadequate stimulation and maternal depression. Evidence based interventions to address these risk factors exist, but often as a separate and overlapping packages delivered through disjointed systems, therefore posing problems in scale-up. A common elements approach based intervention that combines evidence-based elements from packages of care addressing early stimulation, responsive feeding and maternal distress have been developed.

Objectives: The current study aims to develop an online training curriculum to train lay health workers in common elements based intervention to improve maternal psychological well-being and improve mother-infant interaction among distressed mothers in low resource rural community settings of Pakistan. The impact of intervention on maternal well-being, infant growth, nutrition and development will be evaluated at 12-months post-partum.

Method: A two arm, single blind, individual randomized controlled trial (RCT) will be carried out in the community settings of the rural sub-district of Gujar Khan in Rawalpindi, Pakistan. 250 Pregnant women in third trimester of pregnancy, screened positive for psychological distress on Self-Reporting Questionnaire (SRQ), cut-off score ≥ 9, will be randomized on 1:1 allocation ratio into intervention (n=125) and Treatment as Usual (TAU) arms (n=125). The participants in the intervention arm will receive 15 monthly sessions of intervention by community volunteers at home. First three sessions will be delivered in the third trimester of pregnancy followed by one monthly session for 12 months. The primary outcome will be caregiver-infant interaction at 12-months post-partum. The maternal secondary outcomes include maternal psychological wellbeing, quality of life, social support and empowerment. Maternal outcomes will be measured at baseline, 6-months and 12-months post-partum. Infant secondary outcomes include growth, nutrition and development and will be measured at 12 months. A mixed-methods process monitoring and evaluation will be conducted to inform the feasibility of intervention delivery.

Discussion: The outcomes of the study will be a common-elements based online training curriculum for training of community volunteers in intervention to improve maternal psychological well-being and mother-infant interaction in low resource rural community settings at-scale.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with third trimester (28 gestational week)
* Age 18-40 years
* Intent to reside in the study areas until the completion of the study
* Score ≥9 on the SRQ

Exclusion Criteria:

* Women who require immediate or on-going medical or psychiatric care reported.
* Severe previous or current obstetric morbidity including eclampsia and antepartum hemorrhage;
* Medical disorders that require inpatient management (e.g., diabetes, hypertension, thromboembolism, cardiac disease)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants
Enrollment: 250 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Observation of Mother and Child Interaction Tool (OMCI) | At 12-months postpartum
  Maternal responsive caregiving behaviours will be assessed using the Observation of Mother and Child Interaction (OMCI) tool . OMCI tool is based on responsive parenting framework proposed by Landry and colleagues. The research assistants will observe a live 5-minute mother-infant interaction while mother and infant will play together with a picture book. The tool comprises of 19 items covering maternal affect, maternal touch, maternal verbalization, sensitivity and contingent responses, scaffolding, language stimulation, focus, child affect, child focus, child's communication efforts, and mutual enjoyment. The scoring format is based on the frequency of the occurrence of behaviours with higher scores indicating more responsive interactions. The OMCI tool has been validated for use in similar population in Pakistan.

SECONDARY OUTCOMES:
Bayley's Scales of Infant Development (BSID III) | At 12-months postpartum
  Bayley's Scales of Infant Development (BSID III) will be used to measure cognitive, language, motor, socio-emotional development and adaptive behaviours. Each item is rated on 0 or 1. Higher scores indicate better development and functioning.
Ages and Stages Questionnaire 3rd Edition (ASQ3) | At 12-months postpartum
  Ages and Stages Questionnaire 3rd Edition (ASQ3) will be used to measure developmental delays in communication, gross motor, fine motor, problem solving, and personal social domains. It provides cut-off score in 5 domains of development that indicates possible need for further evaluation. It highlights results that fall in a "monitoring zone," to make it easier to keep track of children at risk. Items are rated on 3-point likert scale, yes (10), sometime (5) and not yet (0). Higher score indicates that child is developing well.
The Home Observation for Measurement of the Environment Scale (HOME) | At 12-months postpartum
  Quality and quantity of stimulation and support in the child's home will be measured using home inventory. It has 45 items, rated on dichotomous scale, yes (1) or no (0). It has six sub-scales including parental responsiveness, acceptance of child, organization of environment, learning materials, parental involvement, variety in experience. Higher score shows more enriched home environment.
Anthropometric measurements | At 12-months postpartum
  Infants in both groups will be weighed and measured with standard techniques. Growth data will be converted into SDs (Z scores) for weight and length with Epi Info 2002 (version 3.4.1).
Early breastfeeding (EBF) scale | At 6-months postpartum
  Assessors will document what the infant was fed in the last 24 hours at 6 months postpartum. This information will be categorized as either EBF, partial breastfeeding (giving an infant some breastfeeding, and some artificial foods, either milk, cereal, or other food items), or no breastfeeding, using three items scale. The items will be rated on 3-point likert scale; yes (1), no (0) and don't know (888). Lower score represents that infant is not exclusively breastfed. If the infant will not exclusively breastfeed, details of when (age of infant) and why EBF was discontinued will be recorded. At the first follow-up immediately after delivery, details about early initiation, discarding colostrum, use of pre-lacteals, and reasons for delaying or not initiating breastfeeding will be assessed۔
Number of diarrhoeal episodes | At 6 and 12-months postpartum
  The number of diarrhoeal episodes in the infants during the 2 weeks before interview will be recorded at 6 and 12 months post-partum, with a questionnaire used in previous studies. Diarrhoea will be defined as three or more unformed stools passed in 24 h, and a diarrhoeal episode will be defined as being separated from another episode by at least 3 diarrhoea-free days.
Immunization record form | At 6 and 12-months postpartum
  Records of immunization will be assessed for all infants in the study, and infants will be classified as those with or without up-to-date immunisation status 6 and 12 months postpartum.
Self-Reporting Questionnaire (SRQ) | At baseline, 6 and 12-months postpartum
  Maternal distress will be measured by the Self Reporting Questionnaire (SRQ). SRQ is a 20-item self-report measure to detect non-specific psychological distress, developed by the World Health Organization. The SRQ items are scored 0 or 1. A score of 1 indicates the presence of symptoms of psychological distress during past month and a score of 0 indicates absence of symptoms. The maximum score indicates presence of higher psychological distress.
Pediatric Quality of Life Inventory (PedsQL) | At baseline and 12-months postpartum
  Caregivers' health related quality of life will be measured by Paediatric Quality of Life Inventory (PedsQL) family impact module. The PedsQL is 36 item impact module scale that encompasses 6 sub-scales measuring parent self-reported functioning. These subscales measure physical functioning, emotional functioning, social functioning, daily activities and family relationships. Items are rated on a 5-point Likert scale (0 = never to 4 = almost always). Higher scores indicate better functioning
Multi-Dimensional Scale of Perceived Social Support (MSPSS) | At baseline and 12-months postpartum
  The level of social support will be measured using Multi-Dimensional Scale of Perceived Social Support (MSPSS). It includes 12 items which cover three dimensions: support from family, friends and significant other. Each item is rated on a 7-point Likert-scale (1 = very strongly disagree; 7 = very strongly agree). A total score is calculated by summing the responses of all items (range 12-84) with higher scores indicating higher levels of perceived social support.
World Health Organization Disability Assessment Schedule (WHODAS-12) | At baseline and 12-months' post-partum
  Caregiver's level of functioning will be measured using World Health Organization Disability Assessment Schedule (WHODAS-12). WHODAS assesses participants' health-related difficulties in the level of functioning in six domains of life (understanding and communicating; moving and getting around; attending to one's hygiene, dressing, eating and staying alone; interacting with other people; domestic responsibilities, leisure, work and school and joining in community activities, participating in society) over the past 30 days. It has 12 items rated on 5-point likert scale, 1 to 5. High score represents more disability/ impaired functioning.
Maternal Financial Empowerment Scale | At baseline and 12-months' post-partum
  Women's empowerment will be measured using a questionnaire consisting of: (a) two items previously used in the same population that assess financial empowerment (i.e., whether a woman is given a lump-sum of money for day-to-day expenses and whether she can make independent decisions about its use) and (b) 7 items to measure relative freedom from domination within the family (i.e., whether in the past year family had taken money, land, jewellery or livestock from her against her will, prevented her from visiting her parental home, or prevented her from working outside the home) and economic security and contribution (i.e., does she possess any land, productive assets, and or cash). Women who answer 'yes' to both items on financial empowerment and three items from economic security and contribution subscales and 'no' to all items regarding family domination will be classified as 'empowered'.
Client Service Receipt Inventory (CSRI) | At baseline and 12-months postpartum
  Utilization of health care will be measured by Client Service Receipt Inventory (CSRI) adapted for perinatal population of Pakistan. It measures participants' use of health and social care services, accommodation and living situation, family income and social benefits. The data collected through the CSRI can be used to calculate service costs and total costs of care for each research participant.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Usman Hamdani, PhD, Principal Investigator — Human Development Research Foundation, Pakistan
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available along with the study protocol.
Supporting Information: Study Protocol
Time Frame: The data will be available beginning 9 months and ending 36 months following article publication.
Access Criteria: The data will be shared with investigators who provide a methodologically sound proposal and state that data will be used for purpose of individual participant data meta-analysis only. The research proposals should be directed to syedusmanhamdani@gmail.com to gain access of the data. The data requestors will need to sign a data access agreement as well.

REFERENCES:
- [Background] Rasheed MA, Yousafzai AK. The development and reliability of an observational tool for assessing mother-child interactions in field studies- experience from Pakistan. Child Care Health Dev. 2015 Nov;41(6):1161-71. doi: 10.1111/cch.12287. Epub 2015 Sep 9. PMID 26350208
- [Background] Albers CA, Grieve AJ. Test review: Bayley, N.(2006). Bayley scales of infant and toddler development-third edition. San Antonio, TX: Harcourt assessment. Journal of Psychoeducational Assessment. 2007;25(2):180-90.
- [Background] Squires J, Bricker DD, Twombly E. Ages & stages questionnaires: Paul H. Brookes Baltimore, MD; 2009.
- [Background] Caldwell BM, Bradley RH. Home observation for measurement of the environment: University of Arkansas at Little Rock Little Rock; 1984
- [Background] Committee WE. Physical status: the use and interpretation of anthropometry. http://helid digicollection Org/en/d/Jh0211e/. 1995.
- [Background] Sikander S, Maselko J, Zafar S, Haq Z, Ahmad I, Ahmad M, Hafeez A, Rahman A. Cognitive-behavioral counseling for exclusive breastfeeding in rural pediatrics: a cluster RCT. Pediatrics. 2015 Feb;135(2):e424-31. doi: 10.1542/peds.2014-1628. Epub 2015 Jan 12. PMID 25583916
- [Background] Beusenberg M, Orley JH, Organization WH. A User's guide to the self reporting questionnaire (SRQ. Geneva: World Health Organization; 1994.
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Zimet GD, Dahlem NW, Zimet SG, Farley GKJJopa. The multidimensional scale of perceived social support. 1988;52(1):30-41.
- [Background] Üstün TB, Kostanjsek N, Chatterji S, Rehm J. Measuring health and disability: Manual for WHO disability assessment schedule WHODAS 2.0: World Health Organization; 2010.
- [Background] Rahman A, Sikander S, Malik A, Ahmed I, Tomenson B, Creed F. Effective treatment of perinatal depression for women in debt and lacking financial empowerment in a low-income country. Br J Psychiatry. 2012 Dec;201(6):451-7. doi: 10.1192/bjp.bp.112.109207. Epub 2012 Nov 8. PMID 23137731
- [Derived] Huma ZE, Gillani A, Shafique F, Rashid A, Mahjabeen B, Javed H, Wang D, Rahman A, Hamdani SU. Evaluating the impact of a common elements-based intervention to improve maternal psychological well-being and mother-infant interaction in rural Pakistan: study protocol for a randomised controlled trial. BMJ Open. 2021 Jul 7;11(7):e047609. doi: 10.1136/bmjopen-2020-047609. PMID 34233989